CLINICAL TRIAL: NCT04099160
Title: Cross-cultural Adaptation of Revised Neurophysiology of Pain Questionnaire Into Turkish Language
Brief Title: Turkish Version of Revised Neurophysiology of Pain Questionnaire
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hatice Gül, Principal Investigator, Akdeniz University
Other Study IDs: 34878437-199-E.115170
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Chronic Low-back Pain; Neck Pain
Keywords: neurophysiology pain questionnaire; reliability; validity; pain; low back pain
MeSH Terms: conditions — Neck Pain; Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation — The Turkish version of the Revised Neurophysiology of Pain Questionnaire will be applied to patients with chronic spinal pain at the beginning of the study and a week later. The Visual Analogue Scale and the Short Form-36 (SF-36) questionnaire will be applied to patients only at the beginning of the stuy.

SUMMARY:
The Neurophysiology of Pain Questionnaire was first developed in English to test whether healthcare staff and patients could exactly understand pain neurophysiology. This questionnaire which contains 19 items was developed from the exam questions of students interested in post-graduate pain medicine. Catley et al. (2013) investigated the psychometric properties of the modified Neurophysiology of Pain Questionnaire with a few word differences from the original version by conducting a rash analysis on 300 patients with chronic spinal pain. Acceptable internal consistency and test-retest reliability of the questionnaire were recorded. However, it was stated that 7 items negatively affect psychometric properties of the questionnaire. As a result, the author concluded that the questionnaire had sufficient psychometric properties for use in chronic spinal pain subjects, but further studies were needed. The Neurophysiology of Pain Questionnaire was used to measure a knowledge about pain in different studies. The validity and reliability studies of the Dutch, French and Brazlian Portuguese versions of the Neurophysiology of Pain Questionnaire were conducted in the literature. The aim of our study was to translate the Revised Neurophysiology of Pain Questionnaire into Turkish language and to investigate its psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal pain lasting more than three months
* Patients who older than 18 years of age
* Patients who can understand and read Turkish.

Exclusion Criteria:

* Patients with specific spinal pain such as trauma, fracture, infection, inflammatory disease and tumor
* Patients who have undergone spinal surgery in the last 3 months
* Patients who have received pain neurophysiology education in the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic spinal pain
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
The Revised Neurophysiology of Pain Questionnaire | Two minute
  The Revised Neurophysiology of Pain Questionnaire consists of 12 items and measuring the level of knowledge about pain neurophysiology. High score indicates a high level of knowledge about pain neurophysiology.

SECONDARY OUTCOMES:
Visual Analogue Scale | 1 minute
  Visual Analogue Scale assessed pain severity. Visual Analog Scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of pain. hence the left end is usually labeled 'no pain', and the right end usually labeled 'extreme pain'. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark by using a ruler. The scale is provided a range of scores from 0-100. High score indicates a high level of pain..
Short Form-36 | Ten minute
  Short Form-36 (SF-36) questionnaire has 8 subscales such as physical function, role limitations due to physical problems, pain, general perception of health, energy, social function, role limitations due to emotional problems, mental health. This questioonaire evaluate quality of life. Scales have a fairly small range of response options, and scores are multiplied up to 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Gül, Ph.D, Principal Investigator — Akdeniz University
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz University Department of phyiotherapy, Antalya
  - Akdeniz University Medical Ethics Committe, Antalya

IPD SHARING:
Plan to Share IPD: No
The data obtained from patients at the beginning and a week later will be analyzed with SPSS program.

REFERENCES:
- [Background] Catley MJ, O'Connell NE, Moseley GL. How good is the neurophysiology of pain questionnaire? A Rasch analysis of psychometric properties. J Pain. 2013 Aug;14(8):818-27. doi: 10.1016/j.jpain.2013.02.008. Epub 2013 May 4. PMID 23651882